CLINICAL TRIAL: NCT03953976
Title: INRT- AIR: A Prospective Phase II Study of Involved Nodal Radiation Therapy Using Artificial Intelligence-Based Radiomics for Head and Neck Squamous Cell Carcinoma
Brief Title: INRT-AIR: A Prospective Phase II Study of Involved Nodal Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2019-0711
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET-CT at 3 months and ENT evaluation (Experimental): Treatment to the gross primary and nodal disease (70 Gy), with suspicious nodes treated to 66.5 Gy, all in 35 fractions. CT and PET-CT are required for nodal assessment. Restaging PET-CT must be performed between 11-14 weeks from the completion of treatment. The patient must see an otolaryngologist after the PET-CT to decide on post-treatment neck dissection per the surgeon's judgement. Patients will then be seen every 3 months (+/- 2 weeks) for the first year, and then at least every 6 months (+/-2 weeks) until the 36 month. Subsequent and intervening follow-up visits will be made per physician preference
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy (IMRT) — Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel). 6.5-7 weeks of radiotherapy or chemoradiotherapy

SUMMARY:
Elective nodal irradiation has been a longstanding standard-of-care in the management of mucosal squamous cell carcinoma of the head and neck. Recent studies have suggested that reduced elective dose and volume may be a viable approach to improve toxicity. In this study, we are eliminating the elective neck treatment, focusing therapy on involved and suspicious nodes.

DETAILED DESCRIPTION:
We recently completed and reported a successful study (INFIELD) using reduced elective dose (40 Gy) and volume (involved echelons + 1) for oropharynx and larynx cancer. In INRT-AIR (Involved Nodal Radiotherapy using AI-based Radiomics), we are eliminating the elective neck treatment altogether, using radiologic and radiomic-based criteria to focus treatment on the nodes themselves. Eligible patients include previously untreated patients with stage I-IVB oropharynx, larynx and hypopharynx cancer, excluding T1-2 glottic carcinoma. Patients requiring chemotherapy may receive cisplatin, cetuximab, or carboplatin-paclitexel.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-proven diagnosis of squamous cell carcinoma of the oropharynx, larynx, or hypopharynx. Squamous cell carcinoma of unknown primary is not allowed.
2. Patients must have clinically or radiographically evident measureable disease at the primary site and/or nodal stations. Diagnostic lymph node excision (< 2 nodes) is also allowable.
3. Patients may undergo a diagnostic or therapeutic transoral resection for a T1-2 tonsil or base of tongue cancer.
4. Clinical stage I-IVB (AJCC, 7th edition); stages I-II glottic cancer are excluded
5. Age ≥ 18 years.
6. ECOG Performance Status 0-2
7. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   7.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
8. Negative serum pregnancy test within 2 weeks before registration for women of childbearing potential.
9. Neck CT and/or neck MRI, and PET-CT (at least skull-to-thigh).
10. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Distant metastasis.
2. Inability to undergo PET-CT.
3. Stage I and II glottic carcinoma.
4. Gross total excision of both the primary and nodal disease.
5. Synchronous non-skin cancer primaries outside of the oropharynx, larynx, and hypopharynx except for low- and intermediate-risk prostate cancer and synchronous well-differentiated thyroid cancer; in the latter case, surgery may occur before or after treatment, provided all other eligibility criteria are met .
6. Prior invasive malignancy with an expected disease-free interval of less than 3 years.
7. Prior systemic chemotherapy for the study cancer; prior chemotherapy for a remote cancer is allowable
8. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
9. Subjects may not be receiving any other investigational agents.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy agents in this study (if necessary).
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
12. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
13. History of severe immunosuppression, including HIV, and organ or autologous or allogeneic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
To determine the risk of solitary elective volume recurrence following elective volume reduction using INRT. | 2 years
  Definition: solitary means that the recurrence occurred without a preceding or synchronous in-field or distant recurrence

SECONDARY OUTCOMES:
Comparison of SEVR risks by p16 status and anatomic site | 2 years
EORTC QLQ-C30 Summary score | 36 months
  The EORTC QLQ-C30 Summary Score is calculated from the mean of 13 of the 15 QLQ-C30 scales. Patients rate overall health and quality of life.
EORTC QLQ-C30 Physical and role functioning subscales | 36 months
  Patients rate overall health and quality of life.
EORTC HN35 Dry mouth and sticky saliva subscales | 36 months
  Patients report to which extent they experience symptoms or problems during one week.
MDADI global, emotional, functional and physical subscales | 36 months
  Questionnaire asks for views about swallowing ability.
EQ-5D global score (0-100) | 36 months
  Patients describe health for current day regarding mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Grade 3-4 acute and late toxicity | 2 years
  According to NCI's CTCAE v4.0 toxicity criteria
Gastrostomy placement and subsequent removal rate | 2 years
  To estimate the rates gastrostomy dependence at 3, 6, 12 and 24 months following treatment with INRT.
To characterize patient utilities following treatment with INRT. | 2 years
  Average patient utilities (derived from EQ-5D) at baseline, 3, 6, 12, 18, 24 and 36 months from the end of treatment.
To determine 2-year overall and progression-free survival following treatment with INRT | 2 years
  Overall survival (PFS) is defined as the duration of time from start of treatment to time of progression (LR, RR, or DM) or death.
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression (LR, RR, or DM) or death.
To describe the patterns-of-failure following INRT. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David J Sher, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No